CLINICAL TRIAL: NCT02290210
Title: A Placebo-controlled, Randomized, Double-blind, Multicenter Phase 2 Study to Assess the Efficacy and Safety of URC102 in Gout Patients
Brief Title: Phase 2 Study of URC102 to Assess the Efficacy and Safety in Gout Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URC102KR
Record Dates: First submitted 2014-11-04; First posted 2014-11-14 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — URC102

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Placebo (Placebo Comparator): Placebo x 2weeks
  Interventions: Drug: placebo
- URC102 0.25mg (Placebo Comparator): 0.25mg URC102 x 2weeks
  Interventions: Drug: URC102 0.25mg
- URC102 0.5mg (Experimental): 0.5mg URC102 x 2weeks
  Interventions: Drug: URC102 0.5mg
- URC102 1.0mg (Placebo Comparator): 1.0mg URC102 x 2weeks
  Interventions: Drug: URC102 1.0mg
- URC102 2.0mg (Placebo Comparator): 2.0mg URC102 x 2weeks
  Interventions: Drug: URC102 2.0mg

INTERVENTIONS:
Drug: URC102 0.25mg
  Arms: URC102 0.25mg
Drug: URC102 0.5mg
  Arms: URC102 0.5mg
Drug: URC102 1.0mg
  Arms: URC102 1.0mg
Drug: URC102 2.0mg
  Arms: URC102 2.0mg
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety, PK/PD and Urate Lowering Effect of URC102 in gout patients with hyperuricemia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gout

Exclusion Criteria:

* Participated in other clinical study within 12 weeks prior to enrollment, and received an investigational product (including placebo)

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Trend of serum uric acid reduction and trend of serum uric acid levels | weekly for 3weeks
  Frequency of patients with serum uric acid level reduced to < 6.0 mg/dL and < 5.0 mg/dL at each measurement

CONTACTS AND LOCATIONS:
Locations (1):
- JW Pharmaceutical, Seoul, Seocho-dong, South Korea